CLINICAL TRIAL: NCT02595268
Title: A Phase 1, Open-label, Sequential Study to Investigate the Effect of JNJ 63623872 on Pitavastatin in Healthy Subjects
Brief Title: A Study to Investigate the Effect of JNJ-63623872 on Pitavastatin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CR107446; 63623872FLZ1004 (Other: Janssen Research & Development, LLC); 2015-000628-27 (EudraCT Number)
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Healthy; Pitavastatin; JNJ-63623872
MeSH Terms: interventions — pitavastatin; pimodivir

ARMS (1):
- Pitavastatin Then JNJ-63623872 (Experimental): Participants will sequentially receive single oral dose of pitavastatin 1 milligram (mg) on Day 1, followed by JNJ-63623872 600 mg twice daily on Days 4 through 12 with a single oral dose of pitavastatin 1 mg administered in the morning of Day 9. All study drug intakes will be taken orally, under fed conditions (within approximately 10 minutes after completion of a meal).
  Interventions: Drug: Pitavastatin; Drug: JNJ-63623872

INTERVENTIONS:
Drug: Pitavastatin — Participants will receive single oral dose of pitavastatin 1 milligram (mg) on Day 1 and Day 9.
Drug: JNJ-63623872 — Participants will receive JNJ-63623872 600 mg twice daily on Days 4 through 12.

SUMMARY:
The purpose of this study is to evaluate the effect of steady-state concentrations of JNJ-63623872 on the single-dose pharmacokinetics of pitavastatin in healthy participants.

DETAILED DESCRIPTION:
This is a Phase 1, open-label (identity of study drug will be known to participant and study staff), sequential study in healthy volunteers to investigate the potential Pharmacokinetics (PK) effects of JNJ-872 on pitavastatin. The study consists of Screening Phase (28 days), Treatment Phase (Day 1 - Day 12), Follow up (10-14 days and 30-35 days after last study drug intake or drop). The total duration of the study will be approximately 2 months. Participants will sequentially receive the following treatment: a single oral dose of pitavastatin 1 milligram (mg) on Day 1; JNJ-63623872 600 mg twice daily on Days 4 through 12, with a single oral dose of pitavastatin 1 mg administered in the morning of Day 9. All study drug intakes will be taken orally, under fed conditions (within approximately 10 minutes after completion of a meal). Blood samples will be collected to assess pharmacokinetic parameters. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* A female participant of childbearing potential must have a negative serum beta-human chorionic gonadotropin test at Screening and a negative urine pregnancy test on Day -1
* A female participant must agree not to donate eggs (ova, oocytes) throughout the study and for at least 90 days after receiving the last dose of study drug
* A male participant who is sexually active with a woman of childbearing potential must agree to use two effective methods of birth control, and all male participants must also agree not to donate sperm throughout the study and for 90 days after receiving the last dose of study drug
* Participant must have a body mass index (BMI; weight in kg divided by the square of height in meters) of 18.0 to 30.0 kilogram per square meter (kg/m^2), extremes included

Exclusion Criteria:

* Participant has a history of any illness that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant or that could prevent, limit or confound the protocol specified assessments. This may include but is not limited to renal dysfunction [calculated creatinine clearance below 60 milliliter per minute (mL/min) at Screening], significant cardiac, vascular, pulmonary, gastrointestinal (such as significant diarrhea, gastric stasis, or constipation that in the Investigator's opinion could influence drug absorption or bioavailability), endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances, or a predisposition to myopathy
* Participants with one or more laboratory abnormalities as specified in protocol, at Screening as defined by the World Health Organization (WHO) Toxicity Grading Scale
* Participant with a past history of clinically significant heart arrhythmia (extrasystoli, tachycardia at rest) or of risk factors for Torsade de Pointes syndrome (example, hypokalemia, family history of long QT Syndrome)
* Participants with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticaria
* Participants with a history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy witnessed in previous studies with experimental drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Observed Analyte Concentration Just Prior to the Beginning or at the End of a Dosing Interval (Ctrough) of JNJ-63623872 | 72 hour (hr) post-dose on Day 7, 8; predose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16 hr post-dose on Day 9
  Ctrough is the observed analyte concentration just prior to the beginning or at the end of a dosing interval.
Minimum Observed Analyte Concentration (Cmin) of JNJ-63623872 | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16 hr post-dose on Day 9
  Cmin is the minimum observed analyte concentration.
Maximum Observed Analyte Concentration (Cmax) of JNJ-63623872 | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16 hr post-dose on Day 9
  Cmax is the maximum observed analyte concentration.
Time to Reach the Maximum Observed Analyte Concentration (Tmax) of JNJ-63623872 | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16 hr post-dose on Day 9
  Tmax is the actual sampling time to reach the maximum observed analyte Concentration.
Area Under the Plasma Concentration Curve From Time of Administration up to 12 Hours Post Dosing (AUC12h) of JNJ-63623872 | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16 hr post-dose on Day 9
  AUC12h is the AUC from time of administration up to 12 hours post dosing, calculated by linear-linear trapezoidal summation.
Average Steady-state Plasma Concentration (Cavg) of JNJ-63623872 | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16 hr post-dose on Day 9
  Cavg is the average steady-state plasma concentration, calculated by AUC12h / 12 hours at steady-state (12 hours = dosing interval).
Fluctuation Index (FI) of JNJ-63623872 | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16 hr post-dose on Day 9
  Fluctuation index is percentage fluctuation (variation between maximum and minimum concentration at steady-state), calculated as: 100 multiplied by ([Cmax - Cmin] / Cavg).
Observed Analyte Concentration Just Prior to the Beginning or at the End of a Dosing Interval (Ctrough) of Pitavastatin | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16 hr post-dose on Day 1 and Day 9
  Ctrough is the observed analyte concentration just prior to the beginning or at the end of a dosing interval.
Maximum Observed Analyte Concentration (Cmax) of Pitavastatin | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16 hr post-dose on Day 1 and Day 9
  Cmax is the maximum observed analyte concentration.
Time to Reach the Maximum Observed Analyte Concentration (Tmax) of Pitavastatin | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16 hr post-dose on Day 1 and Day 9
  Tmax is the actual sampling time to reach the maximum observed analyte Concentration.
Area Under the Analyte Concentration vs Time Curve (AUC) From Time 0 to the Time of the Last Measurable Concentration (AUClast) of Pitavastatin | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16 hr post-dose on Day 1 and Day 9
  AUClast is the area under the analyte concentration vs. time curve from time 0 to the time of the last measurable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.
AUC From Time 0 to Infinite Time (AUC[0-infinity]) of Pitavastatin | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16 hr post-dose on Day 1 and Day 9
  AUC(0-infinity) is the last observed measurable (non-BQL) concentration; extrapolations of more than 20 percent (%) of the total AUC are reported as approximations.
Apparent Terminal Elimination Rate Constant (Lambda[z]) of Pitavastatin | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16 hr post-dose on Day 1 and Day 9
  Lambda(z) is the apparent terminal elimination rate constant, estimated by linear regression using the terminal log-linear phase of the log transformed concentration vs. time curve.
Apparent Terminal Elimination Half-life of Pitavastatin (T1/2term) | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16 hr post-dose on Day 1 and Day 9
  T1/2term is the apparent terminal elimination half-life, calculated as Lambda(z).
Ratio of Individual Cmax Values Between Test and Reference Treatment (Ratio Cmax,test/ref) of Pitavastatin | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16 hr post-dose on Day 1 and Day 9
  Ratio Cmax,test/ref is the ratio of individual Cmax values between test and reference Treatment. Test is Day 9 (JNJ-63623872 plus pitavastatin) and reference is Day 1(/pitavastatin alone).
Ratio of Individual AUClast Values Between Test and Reference Treatment (Ratio AUClast,test/ref) of Pitavastatin | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16 hr post-dose on Day 1 and Day 9
  Ratio AUClast,test/ref is the ratio of individual AUClast values between test and reference Treatment. Test is Day 9 (JNJ-63623872 plus pitavastatin) and reference is Day 1(/pitavastatin alone).
Ratio of Individual AUC[infinity] Values Between Test and Reference Treatment (Ratio AUC[infinity],test/ref) of Pitavastatin | predose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 16 hr post-dose on Day 1 and Day 9
  Ratio AUC[infinity],test/ref is the ratio of individual AUC[infinity] values between test and reference Treatment. Test is Day 9 (JNJ-63623872 plus pitavastatin) and reference is Day 1(/pitavastatin alone).

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | From Screening up to End of Study (up to 2 months)
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Antwerp, Belgium